CLINICAL TRIAL: NCT05938361
Title: Efficacy of Tildrakizumab in Difficult-to-treat Areas in Psoriasis - ZODIPSO Study
Brief Title: Efficacy of Tildrakizumab in Difficult-to-treat Areas in Psoriasis
Acronym: ZODIPSO
Status: Active, not recruiting | Type: Observational
Sponsor: Clin4all (Network)
Responsible Party: Sponsor
Other Study IDs: 2022-A02735-38
Record Dates: First submitted 2023-05-30; First posted 2023-07-10 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-07

CONDITIONS: Psoriasis Palmaris; Psoriasis Genital; Psoriasis of Scalp; Psoriasis Plantaris; Psoriasis Nail
Keywords: Psoriasis; tildrakizumab; difficult-to-treat areas
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single group: Cohort of patients with difficult-to-treat psoariasis locations on the nail, scalp, genital and/or palmoplantar area.
  Interventions: Other: Psoriasis clinical assessments; Other: Quality of life evaluation; Other: Satisfaction assessment; Other: Pruritus evaluation

INTERVENTIONS:
Other: Psoriasis clinical assessments — Global evaluation of psoriasis and specific evaluation by areas
Other: Quality of life evaluation — DLQI questionnaire at each visit
Other: Satisfaction assessment — Visual analogic scale at W16, W28, W52
Other: Pruritus evaluation — Visual analogic scale at each visit

SUMMARY:
Psoriasis is a chronic inflammatory disease that affects between 2% and 4% of the French population.Some specific localizations are more difficult to manage, such as the scalp, nails, genital region and palmoplantar localizations.

Tildrakizumab, an anti-interleukin-23 (IL-23) monoclonal antibody, has demonstrated efficacy and safety in the treatment of patients with moderate to severe psoriasis.

Real-life data on the efficacy of Tildrakizumab in unselected patients with these difficult-to-treat locations are still limited.

The aim of the ZODIPSO study is to evaluate the efficacy and safety of Tildrakizumab in patients presented difficult to treat locations in psoriasis : nail, scalp, genital and palmoplantar.

The main objective is to assess the overall response and the specific response to Tildrakizumab at these specific areas up to W52.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory disease that affects between 2% and 4% of the French population. Some specific localizations are more difficult to manage, such as the scalp, nails, genital region and palmoplantar localizations. They are reported at least once during the course of psoriatic disease in more than 80%, 50%, 60%, 12% of patients, respectively.

Despite recent progress in the management of the disease, these localizations remain a challenge for psoriasis patients because of their impact on quality of life and the difficulty of treating them.

Tildrakizumab, an anti-interleukin-23 (IL-23) monoclonal antibody, has already demonstrated efficacy and safety in the treatment of patients with moderate to severe psoriasis in two international multicenter randomized clinical trials : reSURFACE 1 and reSURFACE 2. However, real-life data on the efficacy of Tildrakizumab in unselected patients with these difficult-to-treat locations are still limited.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a diagnosis of moderate to severe chronic plaque psoriasis documented in the medical record,
2. Disease diagnosis > 6 months (regardless of severity at diagnosis)
3. Involvement of at least one of the following areas: nails, scalp, genital, palmoplantar (non-pustular)
4. Indication for treatment by IL-23 inhibitor. Tildrakizumab must be the selected IL-23 inhibitor therapy prior to enrolling the patient in the study. Patients who have previously received previous treatment by IL-23 inhibitors may be included.
5. Patient 18 years of age or older at the inclusion visit
6. French social security beneficiary

Exclusion Criteria:

1. Patient unable to comply with study requirements (i.e.complete study questionnaires)
2. Patient who, in the opinion of the investigator, should not participate in the study. This opinion should be documented in the patient's record.
3. Patient included in an interventional clinical trial at inclusion.
4. Vulnerable patient or patient under court protection
5. Patients with known hypersensitivity to IL-23 inhibitors
6. Patients with HIV or active HBV or HCV infection at the time of inclusion
7. Patient with a history of untreated latent tuberculosis or active tuberculosis at inclusion
8. Patient with any other serious active infection present at inclusion that contraindicates IL23 inhibitors use.
9. Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of moderate to severe chronic plaque psoriasis with specific difficult-to-treat locations.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Specific response to Tildrakizumab at W28 | Week 28
  Percentage of response based on specific assessment on target area (75% improvement of the specific score compared to Baseline visit)

SECONDARY OUTCOMES:
Overall response to Tildrakizumab | Each visit (Week16-Week 28-Week 52)
  Percentage of response based on global assessment compared to Baseline visit
Specific response to Tildrakizumab | Week 16, week 28 and week 52
  Percentage of response based on specific assessment by area compared to Baseline Visit
Adverse events | From baseline visit to Week 52
  Describe adverse events throughout follow-up
Evaluation of pruritus under treatment | Each visit (Baseline,Week 16, Week 28, Week 52)
  Variation in visual analogic scale (VAS) value
Evaluation of quality of life under treatement | Each visit (Baseline, Week16, Week 28, Week 52)
  Dermatology Life Quality Index (DLQI) score compared to Baseline Visit
Evaluation of satisfaction under treatement | Each follow-up visit (Week 16, Week 28, Week 52)
  Variation in visual analogic scale (VAS) value

CONTACTS AND LOCATIONS:
Overall Officials: Ines ZARAA, MD, Principal Investigator — Saint Joseph hospital Paris
Locations (1):
- Service de Dermatologie- Hopital Saint Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: No